CLINICAL TRIAL: NCT03589365
Title: Preterm Birth and Long Term Consequences on Myocardial Functions and Structure
Acronym: PREMACOEUR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2017-14
Record Dates: First submitted 2017-08-22; First posted 2018-07-17 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preterm group (Other): young adults born preterm will performed an Magnetic resonance imaging (MRI)
  Interventions: Other: Magnetic resonance imaging (MRI)
- control group (Other): young adults born at term will performed an Magnetic resonance imaging (MRI)
  Interventions: Other: Magnetic resonance imaging (MRI)

INTERVENTIONS:
Other: Magnetic resonance imaging (MRI) — Compare the left ventricular mass of a young adult population born prematurely (Prema group) to that of a group of young adults born at term (Witness group
  The measurements made during this examination are:
  Coronary Reserve Presence of fat in the myocardium Left ventricular mass Left ventricular volume
  The measurements made during this examination are:
  Coronary Reserve Presence of fat in the myocardium Left ventricular mass Left ventricular volume

SUMMARY:
Cardiovascular diseases (hypertension, coronary heart disease, stroke and cardiac insufficiency) are the leading cause of death worldwide. They are a major cause of concern in public health worldwide as well. Their incidence is increasing especially in emerging countries. It has been shown through epidemiological and experimental studies that these cardiovascular diseases are influenced by environmental factors which can act early during different periods of the development. Preterm birth is an emerging risk factor of cardiovascular diseases. Preterm birth rate varies accordingly to countries from 6 % to 14 % and accounts for 80% of low birth weight. These past thirty years have shown an improvement in the management and survival rate of these babies. The number of preterm infants reaching adulthood is thus increasing. Long term effects of preterm birth on cardiovascular diseases are little known.

However, emerging evidence suggest that preterm birth affects certain functions and structure. A significant increase in blood pressure and alterations on the vascular, metabolic, and renal systems have been reported in healthy young adult born preterm. And abnormal heart shape with left ventricular hypertrophy have been demonstrated in these population (Oxford)

DETAILED DESCRIPTION:
Cardiovascular diseases (hypertension, coronary heart disease, stroke and cardiac insufficiency) are the leading cause of death worldwide. They are a major cause of concern in public health worldwide as well. Their incidence is increasing especially in emerging countries. It has been shown through epidemiological and experimental studies that these cardiovascular diseases are influenced by environmental factors which can act early during different periods of the development. Preterm birth is an emerging risk factor of cardiovascular diseases. Preterm birth rate varies accordingly to countries from 6 % to 14 % and accounts for 80% of low birth weight. These past thirty years have shown an improvement in the management and survival rate of these babies. The number of preterm infants reaching adulthood is thus increasing. Long term effects of preterm birth on cardiovascular diseases are little known.

However, emerging evidence suggest that preterm birth affects certain functions and structure. A significant increase in blood pressure and alterations on the vascular, metabolic, and renal systems have been reported in healthy young adult born preterm. And abnormal heart shape with left ventricular hypertrophy have been demonstrated in these population (Oxford) The aims of this study are to evaluate the effects of preterm birth on heart functions and in a cohort of healthy young adults born preterm. Early alterations could be observed, before the onset of disease. This study will include 60 young adults aged from 18 to 30 years, 30 of them born preterm (Preterm group) and 30 born at term with normal birth weight (Control group). The groups will be matched for age and gender and tobacco exposition.

Young adults born preterm who will be included in the study were born and followed-up in the Neonatal Unit, APHM, in Marseille. Data from the Control adult born at term are well known and available (Marseille DOHaD Study, D.Barker (University of Southampton, England) and K.Thornburg (OHSU Portland, USA)).

This study addresses the mechanism underlying the association between cardiovascular diseases and preterm birth, and aims to identify early predictive markers in order to guide long term follow-up of these young adults. The results of this study will help to develop specific and accurate diagnostic tools and to implement preventive nutritional or pharmacological strategies.

ELIGIBILITY:
Inclusion Criteria:

For the subjects of the group "Préma":

* age between 18 and 30 years, registered with the French social security system, And signed an informed consent form for the study
* gestational age at birth below 34 years
* no growth restriction in utero (birth weight for age Gestational superior to the 10th percentile)
* matching to term subjects on sex, tobacco consumption And age
* not participating in other studies

For the subjects of the "Witness" group:

* age between 18 and 30 years, registered with the French social security system, And having participated in the study Marseille DOHaD Study
* gestational age between 37 and 41 SA
* birth weight between 25th and 75th percentile
* Cardiac MRI, complete data

For all patients:

Available growth data (health records) including weights And sizes at birth, then at 4 months, 9 months, 2 years, 6 years and 12 years The investigator should ensure by consulting the "National Biomedical research "that the subject is not in a period of exclusion from Other test.

Exclusion Criteria:Medical history of:

Congenital heart disease Endocrine or chronic renal disease Acquired metabolic disease in childhood Non-idiopathic hypertension Malignant disease Obesity related to a characteristic pathology. Any physical or psychological condition that would jeopardize the participation of the subject in the research protocol.- Pregnancy in progress.

- Contra-indications to the realization of an MRI: pacemaker Heart valve prosthesis Intracranial surgery Possibility of having received metal projectiles (splinters Metallic, bullets, shrapnel, etc.) Working in metals Presence of prostheses claustrophobia

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-07 (Estimated); Primary Completion 2019-07 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Left ventricular mass | 45 minutes
  Left ventricular mass will be determined (in mg/m²) by tracing the endo and epicardial contours, including the papillary muscles, on end-systole images and late diastole images from the base to the apex. Two different observers will carry out all the measures.
Left ventricular volume | 45 minutes
  Left ventricular volume will be determined (in ml) by tracing the endo and epicardial contours, including the papillary muscles, on end-systole images and late diastole images from the base to the apex. Two different observers will carry out all the measures.

CONTACTS AND LOCATIONS:
Overall Officials: EMILIE GARRIDO PRADALIE, Study Director — Assistance Publique Hôpitaux de Marseille